CLINICAL TRIAL: NCT00707187
Title: Randomized, Placebo-Controlled, Double-Blind, Cross-Over Trial of the Efficacy and Safety of IC351 in Female Patients With Raynaud Phenomenon and Female Sexual Dysfunction Secondary to Systemic Sclerosis
Brief Title: Trial of IC351 in Female Scleroderma Patients With Raynaud's and Sexual Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: James R. Seibold, Professor and Director, UMDNJ
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0220013701
Record Dates: First submitted 2008-06-25; First posted 2008-06-30 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; raynaud phenomenon
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Raynaud Disease | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 35 doses of study medication, IC 351 (20 mg) -- crossover to placebo
  Interventions: Drug: Cialis
- 2 (Experimental): 35 placebo pills followed with 35 study medication (20 mg)
  Interventions: Drug: Cialis

INTERVENTIONS:
Drug: Cialis — 35 pills of study medication (20 mg)

SUMMARY:
Purpose of the study is to evaluate the effectiveness and safety of a new investigational dur, IC351. Study is designed to gather information regarding the possible usefulness of IC351 as a treatment of several blood vessel features of scleroderma. This includes Raynaud phenomenon as well as the vaginal dryness and discomfort associated with scleroderma

ELIGIBILITY:
Inclusion Criteria:

* Female with diagnosis of scleroderma
* Stable sexual relationship with male partner or be sexually active
* Raynaud phenomenon at least 6 times per week
* Willing to attempt sexual activity 1/month during study period

Exclusion Criteria:

* Severe internal organ problems related to scleroderma
* Other gynecologic problems
* Serious depression
* Receiving other experimental and Raynaud treatments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-07; Primary Completion 2002-07; Study Completion 2002-07

PRIMARY OUTCOMES:
Number of Raynaud attacks | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UMDNJ, New Brunswick, New Jersey, United States